CLINICAL TRIAL: NCT05742412
Title: Criteria-based Ambulance Management - Video Indexation VS Standard Indexation On Non-selected Emergency Calls
Brief Title: Dispatch of Emergency Call Using Video Streaming Compared With Traditional Telephone Communication
Acronym: CAM-VISION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Denmark Region (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 3436
Record Dates: First submitted 2023-01-13; First posted 2023-02-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Emergency Medical Dispatch Centre; Video Streaming; Emergency Call; Prehospital Emergency Medical Services
Keywords: Emergency Medical Services; Emergency Medical Service Communication Systems; Audiovisual aid

STUDY DESIGN:
Intervention Model Description: Cluster Randomised Clinical Trials
Who Masked: Participant
Masking Description: The emergency caller (patient or bystander) is initially masked to the intervention (video or telephone communication) when initiating the call to the Emergency Medical Dispatch Center (EMDC). Emergency calls are randomly answered by an EMS Dispatcher using either video or telephone (audio-only) communication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention group: EMS dispatcher using video-based communication in emergency calls.
  In the intervention arm, the EMS Dispatchers are requested to use video in all emergency calls during the 4-month study period.
  Interventions: Device: Video streaming (smartphone camera)
- Control Group (Active Comparator): Control group: EMS dispatcher using telephone-only (audio-only) communication in emergency calls.
  In the control arm, the EMS Dispatchers continue using standard telephone communication (usual care).
  Interventions: Device: Telephone (telephone microphone)

INTERVENTIONS:
Device: Video streaming (smartphone camera) — Adding video streaming as a technical adjunct to the otherwise audio-based-only communication during emergency medical dispatch
  Arms: Intervention Group
Device: Telephone (telephone microphone) — Usual care: Audio-based-only communication using telephone during emergency medical dispatch
  Arms: Control Group

SUMMARY:
In the Emergency Medical Dispatch Center, all EMS dispatchers were divided into one of two clusters with 11 EMS dispatchers in each cluster. Because of few clusters, a matched-pair (MP) design was used based on the average proportion of the dispatched level of urgency (highest level of urgency used as primary matching criteria), years of employment and the average duration of emergency calls in a 3-months period (1st of January 2022 - 31st of March 2022) before the implementation of video streaming. Newly employed personnel where matching was not possible were randomly assigned to one of the two clusters. Prior to the study period, video streaming was gradually implemented in the intervention group during a 6-months period (1st of July 2022 - 31st of December 2022).

Using a cluster randomized setup, the aim was to investigate differences in the management of emergency calls (dispatches) when emergency medical service (EMS) dispatchers use video streaming compared with telephone-only (audio-only) communication. All emergency calls will be randomly distributed between the two clusters.

DETAILED DESCRIPTION:
In Denmark, all emergency medical calls are answered by a nurse- or paramedic trained in dispatching emergencies. The EMS dispatcher determines the level of urgency and the type and number of resources to be allocated (e.g., ambulance, physician-manned vehicle and/or physician-manned helicopter (HEMS). The decision-making process is supported by a standardized national criteria-based dispatch tool called Danish Index for Emergency Care (DI). DI is a tool that classifies the patient's main complaint into different symptom groups (chapters) to determine the level of urgency required and which resources to allocate.

As standard, emergency calls are based on telephone-only (audio-only) communication, which might limit the understanding of a complex clinical presentation.

Previous studies suggest that a visualized clinical presentation could aid the EMS dispatchers in their decision-making and dispatch.

The decision on implementing video streaming has been made by the management board of the Prehospital Emergency Medical Services, Central Denmark Region, Denmark. It has been decided to implement video streaming gradually to allow for this cluster randomized study. Because video streaming is a deemed part of the standard operating procedure (SOP), ethical approval from our local ethical committee is waived. After the study period, video streaming will be implemented in the current control group as the decision to use video streaming as SOP has already been decided.

ELIGIBILITY:
Inclusion Criteria:

* Emergency call to the EMS dispatcher in the EMDC
* EMS dispatcher employed in the total study period
* EMS dispatchers with a completed training period (6 weeks total) at the start of the study period

Exclusion Criteria:

* Emergency calls directed to an EMDC physician or technical logistical personnel not using the criteria-based dispatch tool
* non-emergency calls (health care provider requested prehospital transports)
* EMS dispatcher not employed in the total study period
* EMS dispatchers without a completed training period (6 weeks total) at the start of the study period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20539 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
The frequency of dispatches with the highest level of urgency (A-responses) | Continuously stored during the study period (4 months). Data collection from study termination.
  Defined by the dispatch code generated by the computer-aided dispatch software Logis and stored in the EMDC database

SECONDARY OUTCOMES:
The frequency of dispatches with the levels of urgency A, B, C, D and E | Continuously stored during the study period (4 months). Data collection from study termination.
  Defined by the dispatch code generated by the computer-aided dispatch software Logis and stored in the EMDC database graded in 5 levels.
Mortality, 30-day | Data collection 30 days after study termination (31st of May 2023)
  Mortality within 30 days after study inclusion
Number of participants where the levels of urgency are identical when comparing the ambulance to and from the scene | Continuously stored during the study period (4 months). Data collection from study termination.
  The number and proportion of participant where the level of urgency dispatched by the EMS dispatcher (determining the speed of the ambulance transport to the scene) is identical to the level of urgency determined by the EMS provider (determining the speed of the ambulance transport to hospital).
Length of stay at hospital | Data collection 90 days after study termination or until last patient discharged or dead
  Time from initial hospital admission to hospital discharge to home or care facility
The number of participants needing an ICU admission at hospital | Continuously stored during the study period (4 months). Data collection from study termination.
  Number and proportion of patients needing ICU admission during hospital stay
Number of emergency calls where the dispatched level of urgency is changed during the call | Continuously stored during the study period (4 months). Data collection from study termination.
  Number and proportion of emergency medical calls, where the EMS dispatcher change the level of urgency during the emergency medical call.
Number of emergency calls where the allocated resources is changed during the call | Continuously stored during the study period (4 months). Data collection from study termination.
  Change in allocated resources (e.g., number of ambulances, helicopter, physician manned vehicles etc.) during the emergency call compared with the initially allocated resources.
Number of participants readmitted to hospital within 24 hours after a dispatch without hospital admission (lowest level of urgency - response level E) | 24-hours after study termination
  The number and rate of readmission to hospital within 24 hours among emergency medical calls dispatched at lowest level of urgency (response level E) without allocated prehospital resources (patients only provided with an advice from the EMS dispatcher).
Duration of emergency medical calls | Continuously stored during the study period (4 months). Data collection from study termination.
  The duration of the total call time in minutes.
Time from emergency call to dispatch | Continuously stored during the study period (4 months). Data collection from study termination.
  Time (in minutes) from the start of the emergency medical call to the dispatch (allocated resources with a level of urgency) by EMS dispatcher.
On-scene time | Continuously stored during the study period (4 months). Data collection from study termination.
  Time (in minutes) from EMS provider arrival at scene to departure with the patient.

OTHER OUTCOMES:
Number of participants with return-of-spontaneous circulation (ROSC) after cardiac arrest | Continuously stored during the study period (4 months). Data collection from study termination.
  Number of participants achieving ROSC after cardiac arrest in the prehospital or in-hospital phase of treatment
90 days neurological outcome after cardiac arrest measured by the cerebral performance scale (CPC) | Data collection 90 days after study termination (31st of July 2023)
  Among patients surviving cardiac arrest, neurological outcome will be measured by cerebral performance category (CPC) obtained in the in-hospital electronical patient record 90 days after study inclusion. The CPC ranges from 1 to 5. 1 representing intact function and 5 representing brain death. Favorable neurological function is defined as CPC 1 or 2 and an unfavorable function as 3-5
90 days neurological outcome after cardiac arrest measured by the modified Rankin Scale (mRS) | Data collection 90 days after study termination (31st of July 2023)
  Among patients with cardiac arrest, neurological outcome measured by modified Rankin Scale (mRS) obtained in the in-hospital electronical patient record 90 days after study inclusion. The mRS ranges from 0 to 6. 0 representing no symptoms and 6 representing death. Favorable neurological outcome is defined as mRS 0-2.
Number of patients with Stroke or TIA identified by the EMS dispatcher in the EMDC | Continuously stored during the study period (4 months). Data collection from study termination.
  Recognition of stroke or transient ischemic attack (TIA) by the EMS dispatcher based on the criteria-based dispatch reference work (Danish Index, chapter 26 and the subheadings A03, A04 and B06)
Rate of revascularization treatment (intravenous thrombolysis and/or endovascular treatment (EVT)) among patients with acute ischemic stroke | Continuously stored during the study period (4 months). Data collection from study termination.
  Rate of acute stroke treatment (i.v. thrombolysis and/or endovascular treatment (EVT)) among patients with a timely contact to the EMDC (within 3 hours (thrombolysis) and 24 hours (EVT)).
Primary admission to a hospital offering acute stroke treatment | Continuously stored during the study period (4 months). Data collection from study termination.
  Direct admission by ambulance to a hospital offering acute stroke treatment.
Onset-to-treatment times for patients with acute ischemic stroke treated with i.v. thrombolysis and onset-to-groin-puncture for patients treated with EVT. | Continuously stored during the study period (4 months). Data collection from study termination.
  Time from symptom onset (stroke symptoms) to initiated treatment in-hospital with either iv. thrombolysis or EVT.
Lowest level of urgency (response level E) among children (< 15 years of age) | Continuously stored during the study period (4 months). Data collection from study termination.
  Number and proportion of children (< 15 years of age) dispatched lowest level of urgency (not admitted to hospital and only provided with an advice from the EMS dispatcher)
Re-admissions among children (< 15 years of age) to hospital within 24 hours from a prior emergency call dispatched with lowest level of urgency (response level E) | Continuously stored during the study period (4 months). Data collection from study termination.
  Re-admissions to hospital within 24 hours from a prior emergency call among children (< 15 years of age) initially dispatched with lowest level of urgency (response level E only provided an advice from the EMS dispatcher)
All levels of urgency (response level A, B, C, D and E) among children (< 15 years of age) | Continuously stored during the study period (4 months). Data collection from study termination.
  Defined by the dispatch code generated by the computer-aided dispatch software Logis and stored in the EMDC database

CONTACTS AND LOCATIONS:
Overall Officials: Martin F Gude, MD, Principal Investigator — Prehospital Emergency Medical Service, Central Denmark Region, Denmark
Locations (1):
- Prehospital Emegency Medical Service, Central Denmark Region, Denmark, Aarhus N, Central Jutland, Denmark

REFERENCES:
- [Derived] Gude MF, Valentin JB, Meisner-Jensen M, Bohnstedt-Pedersen NH, Dalgaard AK, Vaeggemose U, Blauenfeldt RA. Video Streaming or Telephone Communication During Emergency Medical Services Dispatch Calls: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Jul 1;8(7):e2519020. doi: 10.1001/jamanetworkopen.2025.19020. PMID 40591356

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT05742412/SAP_000.pdf